CLINICAL TRIAL: NCT05352633
Title: Effects of Intensive Systolic Blood Pressure Lowering Treatment on Out-of-office Blood Pressure - an Ancillary Study to Effects of Intensive Systolic Blood Pressure Lowering Treatment in Reducing RIsk of Vascular evenTs (ESPRIT) Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SFLX2021014
Record Dates: First submitted 2022-04-05; First posted 2022-04-29 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Blood Pressure
Keywords: Intense Pressure Lowering Treatment; Out-of-office Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive BP Arm (Experimental): Participants randomized into the Intensive treatment group will have a goal of SBP <120 mmHg. A two- or three-drug regimen should be initiated at randomization for most participants. Drug doses should be increased and/or additional antihypertensive medications should be added at each visit in the intensive treatment group, usually at monthly intervals, until the participant's goal of <120 mmHg has been reached or the local investigator decides no further antihypertensive medications may be added.
  Interventions: Drug: Intensive BP Arm
- Standard BP Arm (Active Comparator): Participants randomized into the Standard treatment group will have a goal of SBP <140 mmHg. It is expected to achieve a SBP of 135-139 mmHg in as many participants as possible. Medication dose titration or addition of another drug is indicated if SBP is ≥160 mmHg at a single visit or is ≥140 mmHg at two consecutive visits. Down titration should be carried out if the SBP is <130 mmHg at a single visit or <135 mmHg at two consecutive visits.
  Interventions: Drug: Standard BP Arm

INTERVENTIONS:
Drug: Intensive BP Arm — Participants in the Intensive BP treatment group have a goal of SBP <120 mmHg. It is recommended to provide long-acting antihypertensive medications, that is once daily, unless other medication delivery frequency is needed. The local investigator may select among the available study antihypertensive medications. Other drugs not supplied by the trial may also be used as the investigator determines appropriate. One or more medications from the following classes of agents will be provided by the study for use in managing participants in both randomization groups to achieve study goals: Angiotension converting enzyme (ACE)-inhibitors;Angiotension receptor blockers (ARBs); Thiazide-type diuretics; Loop diuretics; Potassium-sparing diuretics; Beta-blockers; Calcium channel blockers (CCBs); Direct vasodilators; Alpha1-receptor blockers; Sympatholytics
  Other Names: Control of SBP to <120 mmHg
  Arms: Intensive BP Arm
Drug: Standard BP Arm — Participants in the Standard BP treatment group have a goal of SBP <140 mmHg. The same medications used in the Intensive BP treatment group will be used for the Standard BP treatment group.
  Other Names: Control of SBP to <140 mmHg
  Arms: Standard BP Arm

SUMMARY:
This study aims to evaluate the effect of intensive treatment (a target clinic based systolic blood pressure(BP) <120mmHg) on 24-hour ambulatory blood pressure and home blood pressure, as well as the effect on White-coat uncontrolled hypertension and masked uncontrolled hypertension, compared with standard treatment (a target clinic based systolic BP <140mmHg).

DETAILED DESCRIPTION:
This study aims to evaluate the effect of intensive treatment (a target clinic based systolic BP <120mmHg) on 24-hour ambulatory blood pressure and home blood pressure, as well as the effect on White-coat uncontrolled hypertension and masked uncontrolled hypertension, compared with standard treatment (a target clinic based systolic BP <140mmHg). The population of this study is from an ongoing multi-centre open label clinical trial which evaluated the effect of intensive systolic hypertension treatment on major cardiac events (ESPRIT study). ESPRIT study enrolled patients with high risk of cardiovascular disease, who were aged≥50 years old with a systolic BP≥130 mmHg, and assigned them randomly to intense hypertension group (a target clinic based systolic BP <120mmHg) or standard hypertension group (a target clinic based systolic BP <140mmHg), with a 3-year follow-up, evaluating the effect of intense hypertension treatment on major cardiac events.

From those eligible ones for the trial, the investigators plan to select 710 to participate in this study. During the 2-3 years of follow-up of the main trial, the participants will be monitored using 24-hour ambulatory blood pressure monitoring, meanwhile one-week home blood pressure monitoring will also be conducted. The two monitoring approaches will be performed twice; once every half year, based on which this study will evaluate the effect of intensive hypertension treatment on 24-hour ambulatory blood pressure and home blood pressure, as well as the effect on White-coat uncontrolled hypertension and masked uncontrolled hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. eligible for the follow up of the main study;
2. content to participate in the sub-study.

Exclusion Criteria:

1. frequently working during night-time;
2. the non - dominant arm could not wear 24-hour ambulatory blood pressure monitoring due to radiation therapy or physical impairment;
3. keep engaged in out-door activities of high physical intensity, e.g. farming or porter, etc.;
4. life expectancy is less than 1 year; such as diagnosed with heart failure, cancer, or end-stage renal disease;
5. the difference of clinical systolic pressure between upper arms was more than 10 mmHg;
6. unable to use smart-phone to upload family blood pressure monitoring data.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 710 (Estimated)
Dates: Start 2022-07-18 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Differences of the mean blood pressure during daytime | During the 2-3 years of follow-up of the main trial (ESPRIT)
  During the 2-3 years of follow-up of the main trial, to compare the differences of the mean blood pressure during daytime among different intervention groups

SECONDARY OUTCOMES:
Proportion of participants with White-coat uncontrolled hypertension | During the 2-3 years of follow-up of the main trial (ESPRIT)
  During the 2-3 years of follow-up of the main trial, to examine the proportion of participants with White-coat uncontrolled hypertension
Differences of the proportions of participants with White-coat uncontrolled hypertension among different intervention groups | During the 2-3 years of follow-up of the main trial (ESPRIT)
  During the 2-3 years of follow-up of the main trial, to compare the differences of the proportions of participants with White-coat uncontrolled hypertension among different intervention groups
Proportion of participants with Masked uncontrolled hypertension | During the 2-3 years of follow-up of the main trial (ESPRIT)
  During the 2-3 years of follow-up of the main trial, to examine the proportion of participants with Masked uncontrolled hypertension
Differences of the proportions of participants with Masked uncontrolled hypertension among different intervention groups | During the 2-3 years of follow-up of the main trial (ESPRIT)
  During the 2-3 years of follow-up of the main trial, to compare the differences of the proportions of participants with Masked uncontrolled hypertension among different intervention groups
Differences of mean blood pressure during night-time | During the 2-3 years of follow-up of the main trial (ESPRIT)
  During the 2-3 years of follow-up of the main trial, to compare the differences of mean blood pressure during night-time among different intervention groups.
Differences of 24-hour mean blood pressure | During the 2-3 years of follow-up of the main trial (ESPRIT)
  During the 2-3 years of follow-up of the main trial, to compare the differences of 24-hour mean blood pressure among different intervention groups.
Differences of the ratios of night-time and daytime blood pressure | During the 2-3 years of follow-up of the main trial (ESPRIT)
  During the 2-3 years of follow-up of the main trial, to compare the differences of the ratios of night-time and daytime blood pressure among different intervention groups.
Differences of mean systolic blood pressure via home blood pressure monitoring | During the 2-3 years of follow-up of the main trial (ESPRIT)
  During the 2-3 years of follow-up of the main trial, to compare the differences of mean systolic blood pressure via home blood pressure monitoring among different intervention groups.
Compare the consistency of clinic-based blood pressure and out-office blood pressure | During the 2-3 years of follow-up of the main trial (ESPRIT)
  During the 2-3 years of follow-up of the main trial, among participants from different intervention groups (intensive and standard groups), to compare the consistency of clinic-based blood pressure and out-office blood pressure (mean SBP during daytime vs mean home blood pressure )

CONTACTS AND LOCATIONS:
Overall Officials: Jing Li, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China